CLINICAL TRIAL: NCT01900340
Title: Intestinal Glucagon-like Peptide-1 (GLP-1) and the Physiological Role in Eating in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKBB 25/11
Record Dates: First submitted 2012-04-03; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Appetite and General Nutritional Disorders
Keywords: GLP-1; satiation peptides; food intake
MeSH Terms: interventions — Sodium Chloride; exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- iv saline, intraduodenal saline (Placebo Comparator): intravenous infusion of saline plus intraduodenal administration of saline
  Interventions: Dietary Supplement: Saline
- IV exendin(9-39) plus intraduodenal (ID) saline (Active Comparator): intravenous infusion of exendin(9-39) plus intraduodenal administration of saline
  Interventions: Drug: Exendin 9-39
- IV saline, intraduodenal nutrient (Placebo Comparator): intravenous infusion of saline plus intraduodenal administration of nutrient
  Interventions: Dietary Supplement: Saline
- Exendin(9-39) plus ID nutrient (Active Comparator): Exendin(9-39) as intravenous infusion plus intraduodenal nutrient administration
  Interventions: Drug: Exendin(9-39) plus ID nutrient

INTERVENTIONS:
Dietary Supplement: Saline — Intravenous saline infusion and intraduodenal administration of saline via feeding tube
  Arms: iv saline, intraduodenal saline
Drug: Exendin 9-39 — IV exendin(9-39) infusion and intraduodenal administration of saline via feeding tube
  Arms: IV exendin(9-39) plus intraduodenal (ID) saline
Dietary Supplement: Saline — IV saline infusion and intraduodenal administration of nutrients
  Arms: IV saline, intraduodenal nutrient
Drug: Exendin(9-39) plus ID nutrient — Exendin(9-39) as intravenous infusion plus intraduodenal nutrient administration
  Arms: Exendin(9-39) plus ID nutrient

SUMMARY:
The aim is to further establish a physiological role for GLP-1 as an endogenous satiety signal by examining the effect of the specific GLP-1 receptor antagonist exendin (9-39) on appetite and food intake in healthy male subjects.

DETAILED DESCRIPTION:
Understanding the exact mechanisms by which GLP-1 inhibits eating can be crucial in order to convert its anorectic action into useful, safe and effective drugs. So far, it is however not clear to what extent GLP-1 is a hormonal regulator of eating or whether the observed effects are rather a pharmacological phenomenon. By applying classical algorithms from endocrinology several criteria must be fulfilled before a hormone can be considered an endogenous physiological satiety signal. One is that exogenous administration of a selective antagonist should prevent the eating-inhibitory effect of GLP-1. At present, cholecystokinin (CCK) is the only peptide in humans identified to fit these criteria. For intestinal GLP-1, it has not been investigated whether a specific GLP-1 receptor antagonist can block the eating-inhibitory effect in humans. The availability of a specific GLP-1 receptor antagonist, exendin (9-39), now makes it possible to further investigate this pathway. Exendin (9-39), is a powerful tool available for human use to characterize of endogenous GLP-1 as a physiological regulator of different biological functions. The molecule has been used to document that endogenous GLP-1 is an important incretin hormone and a regulator of antro-pyloro-duodenal motility. The role of endogenous GLP-1 in regulating food intake and appetite has, however, not been investigated before.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject with a BMI of 19-25 m2/kg
2. Stable body weight for at least three months
3. Normal eating habits
4. Age between 18 and 45 years
5. Sufficient understanding of the German language
6. Subjects understand the procedures and the risks associated with the study
7. Participants must be willing to adhere to the protocol and sign the consent form

Exclusion Criteria:

1. Participation in another clinical trial (currently or within the last 30 days)
2. Smoking
3. Substance abuse
4. Regular intake of medications (except for oral contraceptives)
5. Chronic or acute medical condition including clinically relevant abnormality in physical exam or laboratory values
6. History of gastrointestinal disorders
7. Food allergies

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effect of exendin(9-39)on total calorie intake | 60 min test meal
Effect of exendin(9-39) on total fluid intake | 60 min test meal
Effect of exendin(9-39)on meal duration during an ad libitum test meal. | 60 min test meal

SECONDARY OUTCOMES:
Effect of exendin(9-39)on plasma concentration of glucose | 4 hours blood sampling
Effect of exendin(9-39)on plasma concentration of insulin. | 4 hours blood sampling
Effect of exendin(9-39)on plasma concentration of glucagon. | 4 hours blood sampling
Effect of exendin(9-39)on plasma concentration of GLP-1. | 4 hours blood sampling
Effect of exendin(9-39)on plasma concentration of peptide tyrosine tyrosine (PYY). | 4 hours blood sampling
Effect of exendin(9-39)on plasma concentration of CCK. | 4 hours blood sampling
Effect of exendin(9-39)on plasma concentration of ghrelin. | 4 hours blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital Basel, Phase 1 Research Unit, Basel Switzerland
Locations (1):
- University Hospital Basel, Phase 1 Research Unit, Basel, Switzerland

REFERENCES:
- [Derived] Steinert RE, Schirra J, Meyer-Gerspach AC, Kienle P, Fischer H, Schulte F, Goeke B, Beglinger C. Effect of glucagon-like peptide-1 receptor antagonism on appetite and food intake in healthy men. Am J Clin Nutr. 2014 Aug;100(2):514-23. doi: 10.3945/ajcn.114.083246. Epub 2014 Jun 25. PMID 24965303